CLINICAL TRIAL: NCT06281678
Title: A Phase 2, Open-label, Multicenter Study of IBI363 (PD1-IL2m) in Subjects with Advanced Solid Malignancies
Brief Title: A Study of IBI363 in Subjects with Advanced Solid Malignancies
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI363A202
Record Dates: First submitted 2024-02-04; First posted 2024-02-28 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Melanoma; Non-small Cell Lung Cancer; Colorectal Cancer; Renal Cell Cancer
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- IBI363 (Experimental): IBI363 will be administered as an intravenous (IV) infusion every 2 weeks or every 3 weeks.
  Interventions: Drug: IBI363

INTERVENTIONS:
Drug: IBI363 — IBI363 will be administered as an intravenous (IV) infusion every 2 weeks or every 3 weeks. Subjects will receive study medication until disease progression, toxicity intolerance, withdrawal of consent, the duration of treatment reaches 24 months, or any other reason that requires discontinuation of the study treatment, whichever occurs first.

SUMMARY:
This is a Phase 2, open-label, multicenter study designed to evaluate the efficacy, safety and tolerability of IBI363 (study drug) in subjects with advanced, refractory solid malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects have the ability to understand and give written informed consent for participation in this trial, including all evaluations and procedures as specified by this protocol;
2. Male or female subjects ≥ 18 years old;
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1;
4. Anticipated life expectancy of ≥ 3 months;

Exclusion Criteria:

1. Inadequate bone marrow and organ function;
2. Received previous anti-tumor therapy: Any chemotherapy or targeted small molecule therapy (standard or investigational) within 2 weeks or 5 plasma half-lives. Received Nitrosoureas and mitomycin C within 6 weeks prior to first dose of study drug and during study; Any anti-cancer monoclonal antibody (mAb) within 4 weeks prior to first dose
3. Received live vaccines within 28 days prior to first administration of the study drug or plan on receiving any live vaccine during the study;
4. Has adverse reactions resulting from previous antitumor therapies, which have not resolved to Grade 0 or 1 toxicity according to NCI-CTCAE v5.0 (except for alopecia, fatigue, pigmentation and other conditions with no safety risk according to investigator' discretion) or baseline prior to the first dose of the study drug;
5. Undergone major surgery (Craniotomy, thoracotomy or laparotomy, and other surgery according to investigator' discretion, excluding needle biopsy) within 4 weeks prior to the first dose of the study drug, or who are expected to undergo major surgery during the study period, or who have severe unhealed wounds, trauma, ulcers, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 2 years

SECONDARY OUTCOMES:
Adverse Event （AE） | Up to 90 days post last dose
Dose-limiting Toxicity （DLT） | The DLT observation period is 35 days starting from the first day of cycle 1 (C1D1) for subjects assigned to 1000 μg/kg Q2W, while 28 days starting from the C1D1 for subjects assigned to 2000/3000/4000 μg/kg Q3W.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of California, San Francisco (UCSF), San Francisco, California
  - Ocala Oncology Center, Ocala, Florida
  - BRCR Medical Center, Plantation, Florida
  - University of Kansas Medical Center (KUMC), Fairway, Kansas
  - Michigan Hematology & Oncology Consultants - MedOnc Dearborn, Dearborn, Michigan
  - Michigan Hematology & Oncology Consultants - MedOnc Troy, Troy, Michigan
  - MD Anderson Cancer Center-University of Texas, Houston, Texas
  - Oncology Consultants P.A., Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No